CLINICAL TRIAL: NCT00736190
Title: A Phase IV Study to Evaluate the Efficacy, Safety and Tolerability of Tenofovir DF in Asian-American Adults With Chronic Hepatitis B Infection
Brief Title: A Study to Evaluate Tenofovir Disoproxil Fumarate (DF) in Asian-American Adults With Chronic Hepatitis B Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-174-0123
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Results first posted 2011-08-03 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-11

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B; Hepatitis; Tenofovir disoproxil fumarate; Tenofovir DF; Asian-American
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B; Hepatitis | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TDF (Experimental): 300-mg tablet (marketed formulation) taken orally once daily
  Interventions: Drug: Tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate — 300-mg tablet (marketed formulation) taken orally once daily
  Other Names: Viread

SUMMARY:
The purpose of this study is to evaluate the antiviral activity and safety of tenofovir disoproxil fumarate (TDF) in Asian-American adults (self-reported Asian descent, living in the United States) with chronic hepatitis B infection. All participants will receive active treatment with TDF for 48 weeks.

DETAILED DESCRIPTION:
Efficacy of TDF will be evaluated for reductions in serum HBV DNA, changes in liver enzymes, and the generation of antibody to the virus. Safety will be assessed by evaluating adverse events, laboratory abnormalities, and the development of drug resistance mutations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Asian-American, defined as a person of self-reported Asian ancestry who is residing in the United States (US)
* 18 through 75 years of age, inclusive
* Documented chronic HBV infection, defined as positive serum HBsAg =/> 6 months
* HBV DNA =/> 10,000 copies/mL (PCR method)
* ALT > ULN and </= 10 × ULN at screening or within the past 12 months prior to screening
* Willing and able to provide written informed consent
* Negative serum beta-human chorionic gonadotropin (HCG) pregnancy test (females of child-bearing potential)
* Estimated glomerular filtration rate (creatinine clearance) =/> 60 mL/min/1.73m^2 by the Cockcroft-Gault equation
* Adequate hematologic function (absolute neutrophil count =/> 1,500/mm^3; hemoglobin =/> 10.0 g/dL)
* No prior TDF therapy; participants may have taken < 12 weeks of oral anti-HBV therapy, with the last dose =/> 16 weeks prior to screening; participants may have received prior interferon, but must have discontinued interferon therapy =/> 6 months prior to screening

Exclusion Criteria:

Participants who meet any of the following exclusion criteria are not to be enrolled in this study.

* Pregnant women, women who are breast feeding or who believe they may wish to become pregnant during the course of the study.
* Males and females of reproductive potential who are not willing to use an effective method of contraception during the study. For males, condoms should be used and for females, a barrier contraception method should be used in combination with one other form of contraception.
* Decompensated liver disease defined as direct (conjugated) bilirubin > 1.2 X ULN, prothrombin time (PT) > 1.2 X ULN, platelets < 150,000/mm3, or serum albumin < 3.5 g/dL
* Prior history of clinical hepatic decompensation (eg, ascites, jaundice, encephalopathy) or variceal hemorrhage
* Receipt of prior TDF treatment
* Receipt of =/> 12 weeks of oral anti-HBV nucleoside/nucleotide therapy, or receipt of ANY oral anti-HBV treatment < 16 weeks prior to screening
* Receipt of interferon (pegylated or not) therapy within 6 months of the Screening Visit
* alpha-fetoprotein > 50 ng/mL
* Evidence of hepatocellular carcinoma (HCC)
* Co-infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis D virus (HDV)
* History of significant renal disease (eg, nephrotic syndrome, renal dysgenesis, polycystic kidney disease, congenital nephrosis, acute tubular necrosis, other renal disease)
* History of significant bone disease (eg, osteomalacia, chronic osteomyelitis, osteogenesis imperfecta, osteochrondroses, multiple bone fractures)
* Significant cardiovascular, pulmonary or neurological disease
* Evidence of a gastrointestinal malabsorption syndrome that may interfere with absorption of orally administered medications
* History of solid organ or bone marrow transplantation
* Ongoing therapy with any of the following: nephrotoxic agents, competitors of renal excretion (eg, probenecid), systemic chemotherapeutic agents, systemic corticosteroids, Interleukin-2 (IL-2) and other immunomodulating agents, investigational agents (except with the expressed approval of the Sponsor); administration of any of the above medications must be discontinued at least 30 days prior to the Baseline Visit and for the duration of the study period
* Known hypersensitivity to the study drugs, the metabolites, or formulation excipients
* Any other condition (including alcohol or substance abuse) or prior therapy that, in the opinion of the Investigator, would make the participant unsuitable for the study or unable to comply with dosing requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Fountain Valley, California
  - Hacienda Heights, California
  - Los Angeles, California
  - Monterey Park, California
  - Mountain View, California
  - Oakland, California
  - Palo Alto, California
  - San Jose, California
  - Hamden, Connecticut
  - Baltimore, Maryland
  - Laurel, Maryland
  - Silver Spring, Maryland
  - Englewood, New Jersey
  - Brooklyn, New York
  - Flushing, New York
  - New York, New York
  - Philadelphia, Pennsylvania
  - Fairfax, Virginia
  - Falls Church, Virginia
  - Bellevue, Washington

REFERENCES:
- [Derived] Pan CQ, Chan S, Trinh H, Yao A, Bae H, Lou L. Similar efficacy and safety of tenofovir in Asians and non-Asians with chronic hepatitis B. World J Gastroenterol. 2015 May 14;21(18):5524-31. doi: 10.3748/wjg.v21.i18.5524. PMID 25987775
- [Derived] Pan CQ, Trinh H, Yao A, Bae H, Lou L, Chan S; Study 123 Group. Efficacy and safety of tenofovir disoproxil fumarate in Asian-Americans with chronic hepatitis B in community settings. PLoS One. 2014 Mar 4;9(3):e89789. doi: 10.1371/journal.pone.0089789. eCollection 2014. PMID 24594870

RESULTS

PARTICIPANT FLOW:
Groups:
- A: TDF: Tenofovir disoproxil fumarate (TDF) 300 mg by mouth daily
Period: Overall Study
Arm/Group | A: TDF
Started | 90
Completed | 87
Not Completed | 3
Not completed — Pregnancy | 1
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- A: TDF: Tenofovir disoproxil fumarate 300 mg by mouth daily
Arm/Group | A: TDF
Number analyzed (Participants) | 90
Age Continuous [Mean (Standard Deviation); unit: years] | 36.8 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 90
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 90
Ethnicity [Number; unit: Participants]
  Asian-Chinese | 58
  Asian-Korean | 12
  Asian-Vietnamese | 19
  Asian-Cambodian | 1
Hepatitis B virus (HBV) deoxyribonucleic acid (DNA) [Mean (Standard Deviation); unit: log10 copies/mL] — Plasma HBV DNA was analyzed using polymerase chain reaction (PCR) method.
  log10 copies/mL | 7.484 (1.7678)
Hepatitis B e antigen (HBeAg) [Number; unit: Participants] — Blood samples were collected for HBV serology.
  Participants
    Positive | 53
    Negative | 37
Antibody to HBeAg (Anti-HBe) [Number; unit: Participants] — Blood samples were collected for HBV serology.
  Participants
    Positive | 38
    Unknown | 52
Positive Hepatitis B surface antigen (HBsAg) [Number; unit: Participants] — Blood samples were collected for HBV serology.
  Participants | 90
Alanine aminotransferase (ALT); upper limit of normal (ULN) = 34 U/L [Mean (Standard Deviation); unit: U/L] — Blood samples were collected for serum chemistry.
  U/L | 103.5 (149.61)
ALT (Multiples of ULN) [Mean (Standard Deviation); unit: multiples of ULN] — Blood samples were collected for serum chemistry. Multiples are based on ULN of 34 U/L.
  multiples of ULN | 2.628 (3.5698)
ALT [Number; unit: Participants] — Blood samples were collected for serum chemistry. The ULN for ALT was 34 U/L.
  Participants
    >ULN | 67
    <=ULN | 23
HBV genotype [Number; unit: Participants] — Genotypic analysis was conducted at baseline for all participants.
  Participants
    Genotype B | 43
    Genotype C | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) <400 Copies/mL (<69 IU/mL)
Description: Blood samples were collected from study participants for measuring HBV DNA via polymerase chain reaction (PCR) method.
Time Frame: Week 48
Population: The enrolled-and-treated analysis set included participants who were enrolled into the study and received at least one dose of study drug.
Measure: Number; unit: Participants
Groups:
- Tenofovir DF: 300-mg tablet (marketed formulation) taken orally once daily
Arm/Group | Tenofovir DF
Number analyzed (Participants) | 90
Participants | 74

2. Secondary Outcome: Number of Participants With Alanine Aminotransferase (ALT) Normal at Week 48
Description: Number of participants with normal ALT (at or below the upper limit of normal [ULN] for the central laboratory [34 U/L])at Week 48
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Tenofovir DF
Number analyzed (Participants) | 90
Participants | 59

3. Secondary Outcome: Number of Participants With ALT Normalized (Baseline Values > ULN [34 U/L] and <= ULN at a Subsequent Visit) at Week 48
Description: A normal value at Week 48 after having elevated ALT at baseline; normal ALT is defined as being at or below the ULN for the central laboratory (34 U/L)
Time Frame: Week 48
Population: The enrolled-and-treated analysis set included participants who were enrolled into the study, received at least one dose of study drug, and had baseline ALT > ULN (34 U/L).
Measure: Number; unit: participants
Arm/Group | Tenofovir DF
Number analyzed (Participants) | 67
participants | 40

4. Secondary Outcome: Number of Participants With Composite Endpoint of Hepatitis B Virus (HBV) DNA <400 Copies/mL (<69 IU/mL) and Normal ALT at Week 48
Description: Blood samples were collected for evaluating serum chemistry, including determination of ALT, and for measuring HBV DNA via PCR method. Composite endpoints proposed in the protocol included the percentage of participants with HBV DNA < 400 copies/mL (<69 IU/mL) and normal ALT (ALT <= ULN [34 U/L]); and with HBV DNA < 400 copies/mL, normal ALT, and HBeAg loss/seroconversion. Because so few participants lost hepatitis B e antigen (HBeAg) or developed antibody to hepatitis B e antigen (anti-HBe), only the composite endpoint of HBV DNA < 400 copies/mL and normal ALT was analyzed.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Tenofovir DF
Number analyzed (Participants) | 90
Participants | 55

5. Secondary Outcome: Change From Baseline in FibroTest Value
Description: The FibroTest score is used to assess liver fibrosis and is calculated based on a formula including the participant's age and sex and 5 laboratory parameters: alpha 2 macroglobulin, haptoglobin, gamma-glutamyl transferase (GGT), bilirubin, and apolipoprotein A1. Scores can range from 0.00 to 1.00, with higher scores indicating a greater degree of fibrosis.
Time Frame: Baseline and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tenofovir DF
Number analyzed (Participants) | 90
Scores on a scale | -0.006 (0.1024)

6. Secondary Outcome: Number of Participants With HBeAg/Hepatitis B Surface Antigen (HBsAg) Loss and Seroconversion
Description: HBeAg/HBsAg loss is defined for an individual participant as HBeAg+/HBsAg+ at baseline and HBeAg-/HBsAg- at Week 48. HBeAg/HBsAg serocoversion is defined for an individual participant as HBeAg+/HBsAg+ at baseline and HBeAg-/HBsAg- and anti-HBe+/antibody to hepatitis B surface antigen+ (anti-HBs+) at Week 48.
Time Frame: Week 48
Measure: Number; unit: Participants
Arm/Group | Tenofovir DF
Number analyzed (Participants) | 90
Participants
  HBsAg+ at baseline | 90
  HBsAg- at baseline | 0
  HBsAg+ at Week 48 | 88
  HBsAg data missing at Week 48 | 2
  HBeAg+ at baseline | 53
  HBeAg- at baseline | 37
  HBeAg loss by Week 48 | 6
  Anti-HBe+ seroconversion by Week 48 | 6

7. Secondary Outcome: Number of Participants With HBV DNA < 169 Copies/mL (<29 IU/mL) at Week 48
Description: Blood samples from study participants were collected for measuring HBV DNA via PCR method.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Tenofovir DF
Number analyzed (Participants) | 90
Participants | 73

8. Secondary Outcome: Number of Participants With Composite Endpoint of HBV DNA <400 Copies/mL (<69 IU/mL), Normal ALT, and HBeAg Loss
Description: Composite endpoints proposed in the protocol included the percentage of participants with HBV DNA < 400 copies/mL (<69 IU/mL) and normal ALT (ALT <= ULN [34 U/L]); and with HBV DNA < 400 copies/mL, normal ALT, and HBeAg loss/seroconversion. Because so few participants lost HBeAg or seroconverted to anti-HBe, only the composite endpoint of HBV DNA < 400 copies/mL and normal ALT was analyzed.
Time Frame: Week 48
Reporting Status: Not Posted, anticipated posting 2099-01
Measure: Number; unit: Participants

9. Secondary Outcome: Number of Participants With Composite Endpoint of HBV DNA <400 Copies/mL (<69 IU/mL), Normal ALT, and Seroconversion to Anti-HBe
Description: Composite endpoints proposed in the protocol included the percentage of participants with HBV DNA < 400 copies/mL (<69 IU/mL) and normal ALT (ALT <= ULN); and with HBV DNA < 400 copies/mL, normal ALT, and HBeAg loss/seroconversion. Because so few participants lost HBeAg or seroconverted to anti-HBe, only the composite endpoint of HBV DNA < 400 copies/mL and normal ALT was analyzed.
Time Frame: Week 48
Reporting Status: Not Posted, anticipated posting 2099-01
Measure: unit: Participants

10. Secondary Outcome: Summary of Resistance Surveillance for Participants Without Virologic Breakthrough
Description: Serum was collected for HBV resistance surveillance, and sequence analysis of the HBV polymerase was assessed through di-deoxy sequencing of baseline and postbaseline samples.
Time Frame: Week 48
Population: 10 participants received >= 1 dose of study drug, remained viremic (HBV DNA >= 400 copies/mL) after 48 weeks of TDF treatment, had serum sample for testing, and did not have virologic breakthrough (defined as HBV DNA >= 400 copies/mL [confirmed] after having HBV DNA levels < 400 copies/mL and/or 1-log10 increase [confirmed] in HBV DNA above nadir).
Measure: Number; unit: Participants
Arm/Group | Tenofovir DF
Number analyzed (Participants) | 10
Participants
  No changes in HBV pol/RT | 6
  Changes at polymorphic sites | 1
  Changes at conserved sites | 2
  Unable to genotype | 1

11. Secondary Outcome: Summary of Resistance Surveillance for Participants With Virologic Breakthrough
Description: as for outcome 10
Time Frame: Week 48
Population: 2 participants received >= 1 dose of study drug, remained viremic (HBV DNA >= 400 copies/mL) after 48 weeks of TDF treatment, had serum sample for testing, and had virologic breakthrough (defined as HBV DNA >= 400 copies/mL [confirmed] after having HBV DNA levels < 400 copies/mL and/or 1-log10 increase [confirmed] in HBV DNA above nadir).
Measure: Number; unit: Participants
Arm/Group | Tenofovir DF
Number analyzed (Participants) | 2
Participants
  No changes in HBV pol/RT | 2
  Changes at polymorphic sites | 0
  Changes at conserved sites | 0
  Unable to genotype | 0

12. Secondary Outcome: Summary of Resistance Surveillance for Participants Who Discontinued the Study Early
Description: as for outcome 10
Time Frame: Week 48
Population: 2 participants received >= 1 dose of study drug, discontinued TDF treatment after Week 24 with HBV DNA >= 400 copies/mL, and had serum sample for testing.
Measure: Number; unit: Participants
Arm/Group | Tenofovir DF
Number analyzed (Participants) | 2
Participants
  No changes in HBV pol/RT | 1
  Changes at polymorphic sites | 0
  Changes at conserved sites | 0
  Unable to genotype | 1

ADVERSE EVENTS:
Time Frame: 48 weeks + the follow-up off-study medication period (if applicable). Participants who permanently discontinued study drug were to be followed for 24 weeks off treatment or up to initiation of active treatment, whichever occurred first.
Arm/Group | A: TDF
Serious Adverse Events (participants affected / at risk) | 1/90
Other Adverse Events (participants affected / at risk) | 27/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: TDF (N=90)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A: TDF (N=90)
Nasopharyngitis (Infections and infestations) | 6
Nausea (Gastrointestinal disorders) | 5
Weight decreased (Investigations) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
Headache (Nervous system disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators may discuss or publish results (without Gilead's confidential information) after all results have been publicly disclosed by/with consent of Gilead or study has been completed >=2 years. Proposed publication/presentation and destination details must be submitted >=30 days before submission. The investigator agrees to withhold publication or presentation for an additional 60 days in order to obtain patent protection if deemed necessary.